CLINICAL TRIAL: NCT07374042
Title: Ketoanalogue Supplementation for Muscle Protection in CKD 4 and 5 Patients With Moderately Low Protein Diet
Brief Title: Ketoanalogue Supplementation for Muscle Protection in CKD 4 and 5 Patients With Moderately Low Protein Diet (KETO-PROT-ACTION)
Acronym: KETOPROTACTION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2023 ANIORT 2; 2024-516764-29-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Keto Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keto acid analog (Experimental): Current practice + Keto acid analog (1 tablet / 10 kg body weight) Current practice: protein intake target of 0.6 g/kg/d in order to achieve a dietary protein intake of 0.6 to 0.8 g/kg/d (50% animal protein 50 % plant protein) and total energy intake of 25-35 kcal/kg/d.
  Interventions: Drug: Keto Acid
- Control (No Intervention): Current practice: protein intake target of 0.6 g/kg/d in order to achieve a dietary protein intake of 0.6 to 0.8 g/kg/d (50% animal protein 50 % plant protein) and total energy intake of 25-35 kcal/kg/d.

INTERVENTIONS:
Drug: Keto Acid — Keto acid analog Ketosteril (1 tablet / 10 kg body weight)
  Arms: Keto acid analog

SUMMARY:
Chronic kidney disease (CKD) complicates many pathologies and the rapid increase in its prevalence constitutes a major public health concern. Whatever the cause of kidney failure, high protein consumption is a factor of progression to end-stage kidney disease. A low-protein (0.6 g/kg/d) or a very low-protein (0.3 g/kg/d) diet associated with supplementation with amino acids and/or keto acid analogues (KA) slows down renal function deterioration and prolongs the time before dialysis start. Difficulties in strict protein restriction implementation limit its use to a minority of CKD patients and are difficult to implement in real life.

Recently KDOQI guidelines have recommended a dietary protein intake of 0.55 to 0.6 g/kg/d in CKD 3 to 5 non-diabetic patients "metabolically stable" and 0.6 to 0.8 g/kg/d in diabetic patients. However, the International Society of Renal Nutrition and Metabolism and the French guidelines about management of CKD propose to maintain a protein intake between 0.6 and 0.8 g/kg/d for all patients and as near as possible to 0.6 g/kg/d. This is because for a population, a mean value of 0.66 g/kg/d insures that 95% of patients are above 0.55 g/kg/d (the minimum requirement to avoid a negative nitrogen balance).

Experimental studies and few clinical studies suggest a protective effect of KA supplementation on uremic sarcopenia. Interestingly this effect is also observed in patients with a protein intake of 0.6 to 0.8 g/kg/d and with a dose of KA reduced by half compared to the dose used with VLPD. Moreover, in a preliminary study, we found a nephroprotective effect of KA (1 tablet/5kg body weight) in patients with an average dietary protein intake of 0.7 g/kg/d suggesting a specific effect of KA beyond protein restriction.

The hypothesis is therefore that KA treatment (1 tablet/10kg), together with a dietary protein intake between 0.6 and 0.8g/kg/d, prevent muscle mass loss in patients with stages 4 and 5 CKD. If these results were confirmed, this could expand the population that could benefit from KA supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Older than 18 years of age
* Stage 4 or 5 CKD (eGFR with CKD-EPI 2009 creatinine equation < 30 mL/min/m2), whitout renal replacement therapy or kidney transplantation
* Protein intake 0.6-0.8 g/kg/d (estimated with Moroni formula)
* Social security cover
* Written informed consent

Exclusion Criteria:

* Hospitalization in the past 3 months
* Corticosteroids (> 7.5 mg/d), cytotoxic or immunosuppressive drugs
* Severe symptomatic heart (NYHA 3 or 4) or liver failure (Child Pugh B or C)
* Respiratory failure requiring oxygenotherapy
* Ongoing infection, autoimmune disease or cancer
* Pregnant (e.g., positive human chorionic gonadotrophin [HCG] test) or lactating patients
* Risk of pregnancy: any woman who does not fulfil one of the following criteria:

  * post-menopausal (aged > 45 years with amenorrhea for more than 2 years, or of any age with amenorrhea for more than 6 months and an FSH level > 40 mUI / mL)
  * permanent sterilisation (e.g., occlusion/bilateral ligature of the fallopian tubes, hysterectomy, bilateral salpingectomy, bilateral ovariectomy) or constitutional sterility
  * of childbearing age and using an efficient method of contraception, begun at least 28 days before inclusion. Efficient contraception methods are: oral, injectable or implantable hormonal methods intra-uterine devices sterilisation of the male partner if he is the sole partner abstinence, if compatible with the preferred and usual lifestyle of the individual NB: if child bearing potential changes during the study, the woman must start taking one of the efficient methods of contraception as described above.
* Patients with psychiatric or cognitive disorders rendering them unable to give written informed consent
* Patients unwilling to participate in the study
* Hypersensitivity to the active substances in Ketosteril®
* Hypercalcaemia
* Hypophosphatemia
* Patient under a legal protection (curatorship or tutorship)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Appendicular muscle mass measured by DEXA | at 12 months
  measured by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Julien Aniort, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France